CLINICAL TRIAL: NCT02756481
Title: Treatment Patterns of Care for Patients With Atrial Fibrillation In Venezuela
Brief Title: Local Adaptation of Cost Effectiveness Model for Apixaban Atrial Fibrillation Indication - Venezuela
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CV185-333
Record Dates: First submitted 2015-10-09; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Non-Valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NVAF Treatment patterns: Treatment patterns will be collected during the follow-up period. Data will be directly extracted from medical charts of the arrhythmia unit.
  Anticoagulation use will be reported as drug class: Vitamin K antagonist, antiplatelet, nonsteroidal anti-inflammatory drugs. The following data on anticoagulation use will be collected:
  * Type of treatment, start & stop dates, dosage, administration schedule, method of administration, reason for discontinuation if applicable
  * Type of therapy utilized (monotherapy/combination therapy)
  * Total number of therapy changes or switches through the course of treatment
    * Monitoring visit (visits per month) for International normalized ratio (INR) control by Time in Therapeutic Range(cTTR)
    * Routine care (visits per month) by anticoagulation regimen

SUMMARY:
To characterize treatment patterns and healthcare resource utilization among adults diagnosed with non-valvular atrial fibrillation (NVAF) from the private setting in Venezuela.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of AF (incident and prevalent cases)
* Patient with at least 18 years
* Patients enrolment before and during the study period
* Patients treated in Venezuela

Exclusion Criteria:

* Women who were pregnant at any moment during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This observational, non-interventional, retrospective and longitudinal study of NVAF patients in the private sector in Venezuela based on two study samples to be analyzed separately, medical chart review and an electronic database analysis
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Frequency of Hospitalization | approximately 2 years after enrollment
Duration of Hospitalization | approximately 2 years after enrollment
Frequency of Outpatient visits | approximately 2 years after enrollment

SECONDARY OUTCOMES:
Incidence of Cerebrovascular Disease (CVD) | Up to 3 years
Frequency of Hospitalization due to Cerebrovascular Disease (CVD) | Up to 3 years
Duration of Hospitalization due to Cerebrovascular Disease (CVD) | Up to 3 years
Frequency of Outpatient Visits due to Cerebrovascular Disease (CVD) | Up to 3 years
Incidence of Acute Myocardial Infarction (AMI) | Up to 3 years
Frequency of Hospitalization due to Acute Myocardial Infarction (AMI) | Up to 3 years
Duration of Hospitalization due to Acute Myocardial Infarction (AMI) | Up to 3 years
Frequency of Outpatient Visits due to Acute Myocardial Infarction (AMI) | Up to 3 years
Incidence of Systemic Embolism (SE) | Up to 3 years
Frequency of Hospitalization due to Systemic Embolism (SE) | Up to 3 years
Duration of Hospitalization due to Systemic Embolism (SE) | Up to 3 years
Frequency of Outpatient Visits due to Systemic Embolism (SE) | Up to 3 years
Incidence of Gastrointestinal Hemorrhage (GIH) | Up to 3 years
Frequency of Hospitalization due to Gastrointestinal Hemorrhage (GIH) | Up to 3 years
Duration of Hospitalization due to Gastrointestinal Hemorrhage (GIH) | Up to 3 years
Frequency of Outpatient Visits due to Gastrointestinal Hemorrhage (GIH) | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx